CLINICAL TRIAL: NCT05507359
Title: Effect of Topical Application of Clove Gel Versus Benzocaine Gel on Pain Reduction During Application of Simple Dental Procedures in Children: A Randomized Clinical Trial.
Brief Title: Effect of Topical Application of Clove Gel Versus Benzocaine Gel on Pain Reduction During Application of Simple Dental Procedures in Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farah Ihab Ahmed Rahmy El Sharkawy, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Topical Anaesthia
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clove Gel (Experimental): Group 1: a. The heart rate will be measured using the pulse oximeter before topical application of clove gel.
  b. The site where the rubber dam\ matrix band will be applied will be dried, then topically anesthetized with 4.7% (Pain Out Dental Gel, Colgate Palmolive India Ltd, Solan, India) clove gel for 30-60 seconds.
  c. During rubber dam clamp\ matrix band application, the pain will be evaluated using the Sounds, Eyes, Motor scale.
  d. After the rubber dam clamp\ matrix band application, the child will be asked to choose a face from the Wong-Baker FACES pain rating scale to assess subjective pain.
  e. The heart rate will be measured again using the pulse oximeter to evaluate the child's dental anxiety.
  Interventions: Other: clove gel
- Benzocaine Gel (Active Comparator): 1. The heart rate will be measured using the pulse oximeter before topical application of benzocaine gel.
  2. The site where the rubber dam\ matrix band will be applied will be dried, then topically anesthetized with 20% benzocaine gel for 30-60 seconds (Opahl Gel).
  3. During rubber dam clamp\ matrix band application, the pain will be evaluated using the Sounds, Eyes, Motor scale.
  4. After the rubber dam clamp\ matrix band application, the child will be asked to choose a face from the Wong-Baker FACES pain rating scale to assess subjective pain.
  5. The heart rate will be measured again using the pulse oximeter to evaluate the child's dental anxiety.
  Interventions: Other: Benzocaine gel

INTERVENTIONS:
Other: clove gel — 4.7% (Pain Out Dental Gel, Colgate Palmolive India Ltd, Solan, India) clove gel
  Arms: Clove Gel
Other: Benzocaine gel — 20% Benzocaine gel (Opahl gel)
  Arms: Benzocaine Gel

SUMMARY:
This study is aimed to evaluate the effectiveness of the topical application of clove gel versus topical application of 20% benzocaine gel in pain reduction in children undergoing dental treatment (rubber dam or matrix band application).

DETAILED DESCRIPTION:
Pain is an unpleasant sensory and emotional experience that arises from actual or potential tissue damage or described in terms of such damage. In pediatric dentistry, pain sensation is generated by stimuli like the touch of the needle at the time of local anesthetic administration and is not necessarily caused by tissue damage. Poor pain control, anxiety, and fear of the needle might interfere with the acceptance of local anesthesia and lead to inappropriate dental treatment management.

Fear and anxiety are the most common problems in pediatric dentistry. Needle phobias and fear of pain due to needle prick are very common in children, compromising their dental health. Therefore, various methods (pharmacological or non-pharmacological) have been developed to overcome this problem. Topical anesthetics are the gold standard method used to alleviate pain.

In pediatric dentistry, local anesthesia is the most common procedure that can trigger fear and anxiety in children, but it is an essential measure for pain control. Therefore, an alternative for injectable anesthesia is the use of topical anesthetics.

Rubber dam placement is one of the procedures used daily in dental practice. Unfortunately, anxiety is triggered when injectable anesthesia is applied to control the pain during rubber dam placement. Children perceive rubber dam clamp placement as a painful procedure.

Using an effective topical anesthetic can prevent pain, leading to establishing a trust-based and positive relationship between the pediatric dentist and the child, eliminating the child's fears and anxiety, and developing a positive attitude towards future dental treatments.

Herbal medicine is widely used by approximately 75-80% of the world's population as it has no side effects, is cost-effective, and is locally available. According to the World Health Organization (WHO), the use of herbal remedies exceeds conventional drugs by two to three times. Clove (Syzygium aromaticum) is used in daily life for various potential health benefits and has been used to relieve toothache for ages. It contains active constituents such as eugenol, gallic acid, and eugenyl acetate. It has anesthetic, analgesic, anti-inflammatory, antimicrobial, antifungal, antidiabetic, and antithrombotic action. The mechanism involved in analgesic activity is the activation of calcium and chloride channels in ganglionar cells. The analgesic effect of eugenol is due to its ability to inhibit prostaglandins and other inflammatory mediators.

In the US and UK, researchers reported that 80 percent of pediatric dentists consider rubber dam the gold standard of care; therefore, it is used frequently in daily practice. It provides a means to avoid moisture contamination during fissure sealant placement, especially in the lower molars that are more prone to suffer from saliva contamination. The British Society of Pediatric Dentistry recommended rubber dams for various procedures, including pit and fissure sealants.

Clove is equally effective with benzocaine as a topical agent. Clove has many advantages as it is more than five times cheaper than other topical anesthetics, leading to lower dental costs. It can reduce the dose of drugs the patient absorbs and is widely available even in rural areas. It is especially beneficial in developing countries where the use of topical anesthetics is limited by cost and availability. Therefore, clove can replace the widely used benzocaine topical anesthetic allowing more patients worldwide to benefit from a largely available and cheap topical anesthetic, Few studies have investigated topical anesthetic use for purposes other than reducing needle-related pain). Topical anesthesia is effective only on the surface tissues up to a depth of 2-3 mm. A major drawback of 20% Benzocaine gel is being washed away easily by saliva due to lack of adhesion; it does not adequately flow into the subgingival spaces.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-10 years.
* Cooperative children classified with a rating 3 (positive) or 4 (definitely positive) according to Frankl's behavior rating scale.
* Children with deep pits and fissures requiring pits and fissures sealant in lower permanent first molars.
* Children having class II cavities in lower primary second molars indicated for restoration.

Exclusion Criteria:

* Children with any systemic neurological or psychological disorders.
* Children with known allergy to topical or local anesthetic agents or clove.
* Parental refusal of participation.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception during application of rubber dam or matrix band. | 1 day
  It is measured by Wong-Baker pain rating scale Scale from (0-10)

SECONDARY OUTCOMES:
Child behavior during application of rubber dam or matrix band. | 1 day
  It is measured by SEM (Sound, Eye, Motor Scale) Scale from (0-4)
Heart rate during application of rubber dam or matrix band. | 1 day.
  Pulse oximeter. It is a numerical scale measured by Pulse per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nada Wassef, pHD, Study Chair — Pediatric Dentistry department, Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Alqareer, A., Alyahya, A. and Andersson, L. (2006) "The effect of clove and benzocaine versus placebo as topical anesthetics," Journal of Dentistry, 34(10), pp. 747-750. Available at: https://doi.org/10.1016/j.jdent.2006.01.009. Alqareer, A., Alyahya, A. and Andersson, L. (2006) "The effect of clove and benzocaine versus placebo as topical anesthetics," Journal of Dentistry, 34(10), pp. 747-750. Available at: https://doi.org/10.1016/j.jdent.2006.01.009. Havale, R. et al. (2021) "Comparative evaluation of pain perception following topical application of clove oil, betel leaf extract, lignocaine gel, and ice prior to intraoral injection in children aged 6-10 years: a randomized control study," Journal of Dental Anesthesia and Pain Medicine, 21(4), p. 329. Available at: https://doi.org/10.17245/jdapm.2021.21.4.329. Hu, Y.H. et al. (2018) "Postoperative dental morbidity in children following dental treatment under general anesthesia," BMC Oral Health, 18(1), pp. 1-8. Available at: https://doi.org/10.1186/s12903-018-0545-z. Priyatham, S. and Nuvvula, S. (2016) "Intraoral topical anaesthesia in pediatric dentistry: Review," International Journal of Pharma and Bio Sciences, 7(4), pp. B346-B353. Available at: https://doi.org/10.22376/ijpbs.2016.7.4.b346-353. Shindova, M.P., Belcheva-Krivorova, A. and Taralov, Z. (2022) "Pulse Oximetry in Paediatric Dentistry," International Journal on Recent and Innovation Trends in Computing and Communication, 64(2), pp. 202-206. Available at: https://doi.org/10.3897/folmed.64.e69136. Tandon, S. et al. (2018) " Comparative Evaluation of Mucosal Vibrator with Topical Anesthetic Gel to reduce Pain during Administration of Local Anesthesia in Pediatric Patients: An in vivo Study ," International Journal of Clinical Pediatric Dentistry, 11(4), pp. 261-265. Available at: https://doi.org/10.5005/jp-journals-10005-1523. Wambier, L.M. et al. (2018) "A randomized clinical trial evaluating rubber dam clamp pain reduction from a new topical liposomal anesthetic gel," Pediatric Dentistry, 40(3), pp. 190-194. Yıldırım, S., Tokuç, M. and Aydın, M.N. (2020) "The effect of pre-anesthesia with a needle-free system versus topical anesthesia on injection pain of the inferior alveolar nerve block: a randomized clinical trial," Clinical Oral Investigations, 24(12), pp. 4355-4361. Available at: https://doi.org/10.1007/s00784-020-03301-9.